CLINICAL TRIAL: NCT05519605
Title: Bile Duct Drainage After ERCP Failure: EUS-guided Biliary Versus Percutaneous Transhepatic Drainage
Brief Title: Bile Duct Drainage After ERCP Failure: EUS-BD vs PTBD
Acronym: BESTDRAIN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 113346
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2023-12

CONDITIONS: Pancreatic Cancer; Cholangiocarcinoma; Biliary Obstruction
MeSH Terms: conditions — Pancreatic Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 180 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PTBD after failed ERCP: Patients with a distal malignant obstruction undergoing placement of a percutaneous transhepatic biliary drain after failed ERCP.
- EUS-BD after failed ERCP: Patients with a distal malignant obstruction undergoing EUS-guided biliary drainage after failed ERCP.

SUMMARY:
The vast majority of patients with distal biliary, pancreatic head or uncinate process cancer have jaundice caused by distal malignant obstruction (DMO) of the common bile duct. Biliary drainage by Endoscopic Retrograde Cholangiopancreatography (ERCP) with trans-papillary stent placement is the treatment of choice.

ERCP has a failure rate ranging from 12 - 25 percent. Percutaneous transhepatic biliary drainage (PTBD) is the alternative conventional way to drain the biliary tree after ERCP failure, which is related with substantial morbidity (62%) and mortality (17%). Endoscopic ultrasound (EUS)-guided biliary drainage (EUS-BD) is a novel promising drainage modality with reported excellent outcomes in terms of clinical success and complications.

The implementation of EUS-BD besides ERCP and PTBD into Dutch daily clinical practice raises many questions related to performance, costs, QoL, training, implementation and overall oncological treatment success. This structured learning/proctoring program with an additional national registry provides insights into EUS-BD and how to implement EUS-BD in the Dutch standard of care.

DETAILED DESCRIPTION:
The study is designed as a prospective multicenter registry. The data obtained in this study will enable the EUS-BD procedure to progress to larger multicenter and preferably randomized control trials.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Distal malignant CBD obstruction (from ampulla to 1cm distal to the hilum)
* Indication for biliary drainage after failed ERCP-guided biliary drainage

Exclusion Criteria:

* Previous PTBD and/or EUS-BD
* Inability to provide informed consent
* Pregnancy
* American Society of Anesthesiology (ASA) Grade IV-V

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older with a distal malignant obstruction of the common bile duct with failure of drainage by the initial ERCP will be included in this study. Failed biliary drainage is defined as failed common bile duct cannulation during ERCP by an experienced advanced endoscopist (>100 ERCP/year, case load > 500 ERCP).
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Complications of PTBD vs EUS-BD | 180 days
  The primary outcome measure is a composite of severe complications occurring within 180 days following inclusion, analyzed by intention to treat. Complications we score are: bleeding, perforation, biliary leak, biliary peritonitis, abscess, haemobilia, stent occlusion, cholangitis, pancreatitis, anesthesia related complications, severe post-procedural pain, drain/stent dysfunction, cutaneous fistula, stent migration and drain leakage or dislocation.

SECONDARY OUTCOMES:
Technical success of the initial procedure | 180 days
  Defined as: the ability to access and drain the bile duct by placement of a stent/drain.
Clinical success | 180 days
  A post-intervention reduction of bilirubin below 35 umol/L or a significant decline, so that chemotherapy could be administered at the discretion of the oncologist. Serum bilirubin is routinely measured as part of clinical practice after biliary drainage.
Length of hospital stay | 180 days
  Split into total admission days, length of initial admission and total duration of subsequent admissions; an out-patient procedure performed at the hospital is counted as one admission day
Stent/drain patency | 180 days
  Stent/drain patency is measured by the interval (days) between the time of stent placement and stent/drain malfunction or patient death.
Treatment delay | 180 days
  For each severe complication, the treatment team will be asked whether the complication would alter (delay or modify) the pre-existing treatment plan
Time to re-intervention and number of re-interventions | 180 days
Successful training | 180 days
  Successful training defined as significant progress in learning curve calculated by a CUSUM-analysis
Effect of EUS-BD and PTBD on the difficulty of surgery. | 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The dataset used during this study is available from the corresponding author upon reasonable request.